CLINICAL TRIAL: NCT00879736
Title: A Multi-centre, Randomised Trial in Ontario to Evaluate the Efficacy of Talking Health Together T.M. (T.H.T. in Practice), a Communication Education Intervention for Primary Care Patients With Chronic Disease.
Brief Title: A Study of the Effect of Patient Education (Talking Health Together) in Improving Doctor-patient Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Dr. Marie-Therese Lussier (Unknown); Dr. Claude Richard (Unknown)
Responsible Party: AstraZeneca, Astrazeneca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: THT in practice
Record Dates: First submitted 2009-04-08; First posted 2009-04-10 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2010-10

CONDITIONS: Doctor-patient Communication Improvement
Keywords: Doctor-patient communication; Encounters; Patient education training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- THT PACE eLearning module (Active Comparator): The PACE (prepare, ask, check, express) training methodology will be available to patients before their 2nd doctor visit
  Interventions: Behavioral: THT PACE Training
- THT PACE eLearning module & nurse-led workshop training (Active Comparator): THT PACE eLearning and then nurse-led workshop for training on PACE methodology
  Interventions: Behavioral: THT PACE Training
- Usual care (Placebo Comparator): Patients just go to their doctor as they normally would but get some disease specific information in the form of brochures as do intervention arms
  Interventions: Other: placebo

INTERVENTIONS:
Behavioral: THT PACE Training — Patient training
  Arms: THT PACE eLearning module
Behavioral: THT PACE Training — Patient training
  Arms: THT PACE eLearning module & nurse-led workshop training
Other: placebo
  Arms: Usual care

SUMMARY:
This study is being carried out to see if patients make the lifestyle changes or take their medication as instructed by their doctor during their visit as a result of the T.H.T. patient-education training. Proper information exchange between doctors and patients is an important part of quality health care. Although many patients would like more information, they often do not ask for it directly during doctor-patient visits. The patient-training in this study specifically aims at improving patient participation during medical appointments by building communication skills such as requests for information and sharing health concerns with the doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 40 years of age or greater
* Clinical documentation of diagnosis not to target of at least one of the following: Type II Diabetes Mellitus, Hypertension or Hypercholesterolemia
* Receive a prescribed medication for the chronic disease for which they were included in the study

Exclusion Criteria:

* Patients in active phase of cancer treatment (i.e. chemotherapy or radiotherapy at time of study).
* Inability to carry out the encounter with their physician in English without need of assistance
* Uncomfortable using a computer for routine activities such as regular access to the web and e-mail.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact, compared to Usual Care, of training interventions on patients with chronic disease on patient participation in primary care encounters assessed after intervention. | once

SECONDARY OUTCOMES:
physician satisfaction and sense of partnership with the doctor-patient encounter;
patient perception of quality of doctor-patient communication and relationship and patient confidence in own ability to communicate effectively with their doctor; | Twice
patient perception of the management of their chronic disease(s); and patient recall of discussions of lifestyle recommendations and chronic disease medications discussed during the encounter. | Twice

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Marie-Thérèse Lussier, MD, BSc., MSc., FCMFC, Principal Investigator — Université de Montréal
Locations (5):
- Canada (5):
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kitchener-Waterloo, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Oakville, Ontario